CLINICAL TRIAL: NCT00219947
Title: Viral and Host Factors in the Transmission and Pathogenesis of HIV
Status: Terminated | Type: Observational
Why Stopped: Blood drawing protocol for RUH/ADARC. ADARC ceasing operations at RUH
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Other Study IDs: MMA-448
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: HIV Infections
Keywords: HIV Infection; Acute HIV Infection; Primary HIV Infection; Acute Seroconversion Syndrome
MeSH Terms: conditions — HIV Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- high risk: Blood draw from individuals known to be or at high risk for HIV-infection
  Interventions: Other: blood draw
- diagnosed: Blood draw f rom individuals diagnosed with HIV infection
  Interventions: Other: blood draw

INTERVENTIONS:
Other: blood draw — * T cell subset enumeration
  * Serologic reactivity with HIV antigens
  * Viral load assays by bDNA, PCR, or RT-PCR
  * Routine Laboratory assessments (chemistries, liver function tests, hepatitis serology, RPR)
  * HIV-1 Resistance Testing

SUMMARY:
To study the collection of blood from individuals known to be at high risk for HIV-infection or who have been recently infected with HIV.

The data collected are used for diagnostic, prognostic and management decisions as outlined by current HIV-1 Treatment Guidelines.

DETAILED DESCRIPTION:
This phlebotomy protocol permits the collection of blood from individuals known to be at high risk for HIV-infection or who have been recently infected with HIV.

Participants will have from 10 to 60 ml (approximately 1 to 4 tablespoons) of blood drawn for one or all of the following tests:

* T cell subset enumeration
* Serologic reactivity with HIV antigens
* Viral load assays by bDNA, PCR, or RT-PCR
* Routine Laboratory assessments (chemistries, liver function tests, hepatitis serology, RPR)
* HIV-1 Resistance Testing

These data are used for diagnostic, prognostic and management decisions as outlined by current HIV-1 Treatment Guidelines

ELIGIBILITY:
Inclusion Criteria:

recently infected with HIV-1 HIV-1 negative, and at high risk for infection

Exclusion Criteria:

none

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects are either referred by primary health care providers, self-referred, or may be seeking enrollment in other ADARC clinical trials in the NYC area.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2000-07; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Participants are tested for HIV-1 RNA levels, the presence of antibodies to HIV antigens, and T cell subsets | first visit

SECONDARY OUTCOMES:
Data will be used for diagnostic, prognostic and management decisions as outlined by current HIV-1 Treatment | first visit

CONTACTS AND LOCATIONS:
Overall Officials: Martin M Markowitz, MD, Principal Investigator — Rockefeller University
Locations (2):
- United States (2):
  - Aaron Diamond AIDS Research Center (ADARC), New York, New York
  - Rockefeller University Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Aaron Diamond AIDS Research Center — http://www.adarc.org